CLINICAL TRIAL: NCT00115544
Title: An Open-Label Study of the Safety and Clinical Pharmacology of Stanate® in Infants At-Risk for Exchange Transfusion
Brief Title: Safety and Pharmacology of Stanate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Collaborators: National Children's Hospital, Vietnam (Other)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 64,185-06-2W; no grant or contracts
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2016-02

CONDITIONS: Hyperbilirubinemia
Keywords: neonatal; jaundice; hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia; Jaundice | interventions — tin mesoporphyrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): stannsoporfin 0.75mg/kg
  Interventions: Drug: Stanate
- 2 (Experimental): stannsoporfin 1.5mg/kg
  Interventions: Drug: Stanate
- 3 (Placebo Comparator): saline injection
  Interventions: Drug: Stanate

INTERVENTIONS:
Drug: Stanate — Intramuscular injection of stannsoporfin at 0.75 or 1.5mg/kg for treatment of severe hyperbilirubinemia to prevent exchange transfusion

SUMMARY:
The purpose of this study is to evaluate the effect and safety of Stanate (stannsoporfin) in infants who are at risk for an exchange transfusion and meet the criteria of the protocol.

DETAILED DESCRIPTION:
The present study evaluated the relationship between Stanate® dose, drug safety, and efficacy in a non randomised sequential open label cohort design, in 55 patients. Subjects were term and near term infants at medium or high risk of hyperbilirubinemia with TSB levels approaching the threshold for exchange transfusion. The first cohort began at a dose of stannsoporfin 0.75 mg/kg of birth weight intramuscularly. The dose was then increased to 1.5 mg/kg for cohort 2, and saline was given (placebo) for cohort 3. Safety evaluations consisted of hepatic, renal and hematologic clinical laboratory tests along with serial physical examinations. Long term follow up of all patients to age 6 is planned.

ELIGIBILITY:
Inclusion Criteria:

* Term and near-term healthy infants (may be no more than 14 days of age) with excessive hyperbilirubinemia who are at risk for exchange transfusion according to the AAP guidelines of 2004

Exclusion Criteria:

* No parental consent
* Major known congenital anomaly
* Current use of antibiotics, cardio-respiratory instability, abnormal renal function, hepatitis (as related to TORCH infections)
* Phenobarbital use in either child or mother (30 days prior to child's birth)

Ages: 2 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Reduction of serum bilirubin levels; need for exchange transfusion, safety parameters | 30 days with long term f/u

CONTACTS AND LOCATIONS:
Locations (1):
- National hospital of pediatrics, Hanoi, Vietnam